CLINICAL TRIAL: NCT03289806
Title: Study of the Effects of Docosahexaneoic Acid (DHA) on Post-operative Fibrosis of Trabulectomy Blebs in Glaucoma Surgery
Brief Title: Effects of DHA on Post-operative Fibrosis of Trabulectomy Blebs in Glaucoma Surgery
Acronym: DHA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DELAZZER 2016
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Trabulectomy; Deep Sclerectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fibroblasts of Tenon's capsule (surgical waste)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Glaucoma surgery
  Interventions: Procedure: Samples of fibroblasts from Tenon's capsule
- Controls: Strabismus surgery
  Interventions: Procedure: Samples of fibroblasts from Tenon's capsule

INTERVENTIONS:
Procedure: Samples of fibroblasts from Tenon's capsule

SUMMARY:
Post-operative fibrosis of trabulectomy blebs is a major cause of surgical failure leading to a renewed increase in intraocular pressure. The use of anti-metabolites over many years has made it possible to improve success rates for this surgery but these drugs have numerous adverse effects as they are toxic. Alternative therapies are thus necessary, and we believe that DHA could have antifibrotic effects on fibroblasts and could thus improve success rates in this surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing trabulectomy or deep sclerectomy
* Patients informed about the study

Exclusion Criteria:

- Patients who refuse to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for glaucoma or strabismus
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-01-12 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Test of cell viability by MTT (3-[4,5-dimethylthiazol-2-yl]-2,5-diphenyltetrazolium bromide) | At baseline
Test migration ability by video microscopy | At baseline
Test proliferation with immunohistochemistry (Ki67 staining) | At baseline
Analysis of cell cycle in flow cytometry | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France